CLINICAL TRIAL: NCT01182077
Title: A Phase 1, Open Label, Crossover, Drug Interaction Study of the Pharmacokinetics of ASP015K and Midazolam After Separate and Concomitant Administration to Healthy Adult Subjects
Brief Title: A Study to Assess Drug Interaction of ASP015K and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 015K-CL-PK05
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy; Pharmacokinetics of ASP015K and Midazolam
Keywords: ASP015K; midazolam; healthy volunteers
MeSH Terms: interventions — peficitinib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): ASP015K low dose and midazolam followed by ASP015K high dose and midazolam
  Interventions: Drug: ASP015K; Drug: Midazolam
- Group 2 (Experimental): ASP015K high dose and midazolam followed by ASP015K low dose and midazolam
  Interventions: Drug: ASP015K; Drug: Midazolam

INTERVENTIONS:
Drug: ASP015K — Oral
Drug: Midazolam — Oral

SUMMARY:
The objective of the study is to characterize the effect of multiple doses of ASP015K on the pharmacokinetics of a single dose of midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighing at least 45kg and BMI of 18-32 kg/m2, inclusive
* If female, subject is at least 2 years post menopausal or is surgically sterile per documentation provided by a third party medical professional and the subject is not pregnant as documented by a negative serum pregnancy test
* If male, subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy during the study period

Exclusion Criteria:

* History of any clinically significant disorder, disease or malignancy excluding non-melanoma skin cancer
* Recent history (within 6 months) of drug or alcohol abuse or positive urine screen for drugs of abuse/illegal drugs
* Treatment with prescription drugs or complementary and alternative medicines (CAM) within 14 days prior to study drug administration, or over the counter medication within 1 week prior to study drug administration
* A symptomatic, viral, bacterial or fungal infection within 1 week prior to clinic check-in
* Positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg)
* History of the human immunodeficiency virus (HIV) antibody
* Positive tuberculosis (TB) skin test or Quantiferon Gold test
* Vaccinated within the last 30 days prior to study drug administration
* Received an experimental agent within 30 days or five half-lives, whichever is longer, prior to study drug administration
* Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* Absolute neutrophil count (ANC) <2500 cells/mm3

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables assessed through the analysis of blood and urine samples | Days 1-8 and Days 21-27

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Miami, Florida, United States